CLINICAL TRIAL: NCT00885300
Title: Cloxacillin as Prevention of Double Lumen Infection in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Office of Vice Chancellor for research in Shiraz UMS, Shiraz University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3705
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Double Lumen Infection; Hemodialysis
MeSH Terms: interventions — Cloxacillin; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): cloxacillin 100 mg/ml + heparin 1000iu/ml as catheter lock at the end of hemodialysis
  Interventions: Drug: cloxacillin; Drug: heparin
- 2 (Active Comparator): heparin 1000iu/ml as catheter lock at the end of hemodialysis
  Interventions: Drug: heparin

INTERVENTIONS:
Drug: cloxacillin — cloxacillin 100mg/ml as catheter lock at the end of hemodialysis
  Arms: 1
Drug: heparin — heparin 1000iu/ml as catheter lock at the end of hemodialysis

SUMMARY:
The purpose of this study is to investigate whether cloxacillin lock is effective in prevention of double lumen infection.

DETAILED DESCRIPTION:
Double lumen infection is one of the causes of morbidity and mortality in hemodialysis patients. Many strategies used to prevent it and one of them is antibiotic lock. Thus we select chronic hemodialysis patients and divided them into 2 groups. One group received cloxacillin and heparin as catheter lock and the second group received only heparin lock.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis for 3 months
* at least 2 time dialysis/week

Exclusion Criteria:

* active infection
* acute renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
catheter infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: maryam pakfetart, assistant professor, Study Chair — Shiraz nephro-urology research center
Locations (1):
- Shiraz University Hemodialysis Center, Shiraz, Fars, Iran

REFERENCES:
- [Background] Unver S, Atasoyu EM, Evrenkaya TR, Ardic N, Ozyurt M. Risk factors for the infections caused by temporary double-lumen hemodialysis catheters. Arch Med Res. 2006 Apr;37(3):348-52. doi: 10.1016/j.arcmed.2005.07.010. PMID 16513483